CLINICAL TRIAL: NCT00928343
Title: Double Blind Placebo Controlled Dose Ranging Study for the Assessment of Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Single Ascending Subcutaneous and Oral Doses of GLPG0187 in Healthy Subjects.
Brief Title: First-in-Human Single Ascending Subcutaneous (s.c.) Dose and Single Oral Dose of GLPG0187
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos NV
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0187-CL-101
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — GLPG0187

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG0187 (Experimental): Single dose
  Interventions: Drug: GLPG0187
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0187 — Single ascending subcutaneous doses (subcutaneous solution), and single oral dose (oral solution)
  Arms: GLPG0187
Drug: Placebo — Matching subcutaneous or oral placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) subcutaneous and single oral dose of GLPG0187 compared to placebo.

Also, pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0187 after single subcutaneous and oral administration will be evaluated, and, if applicable, the maximum tolerated dose determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m², inclusive

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single subcutaneous and oral dosing | up to day 10 postdose

SECONDARY OUTCOMES:
Pharmacokinetics of single subcutaneous and oral doses | up to 10 days postdose
Exploratory evaluation of S-CTX | up to 24 hrs postdose

CONTACTS AND LOCATIONS:
Overall Officials: Giocondo Lorenzon, PhD, Study Director — Galapagos NV; Eva Vets, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium